CLINICAL TRIAL: NCT01886274
Title: Transcranial Direct Current Stimulation in the Visual Cortex of Migraine Patients: Neurophysiological and Clinical Implications
Brief Title: Does tDCS is Effective in the Prophylactic Treatment of Migraine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Professor, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Migraine_tDCS
Record Dates: First submitted 2013-06-18; First posted 2013-06-25 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Migraine
Keywords: EEG; migraine; pain; phosphene; tDCs; TMS
MeSH Terms: conditions — Migraine Disorders; Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- tDCS (Experimental): The experimental group received tDCS to the occipital cortex in 12 sessions, 3 days per week.
  Interventions: Device: Transcranial direct current stimulation
- control (Sham Comparator): The control group received sham stimulation to the occipital cortex in 12 sessions, 3 days per week.
  Interventions: Device: Transcranial direct current stimulation
- healthy subjects (No Intervention): This group was submitted to one evaluation session of cortical excitability.

INTERVENTIONS:
Device: Transcranial direct current stimulation — tDCS involves application of very low amplitude direct current via surface scalp electrodes. The applied current modifies the transmembrane neuronal potential and thus influences the level of excitability. Depending on the polarity of active electrodes tDCS can increase or decrease the cortical excitability. The cathodal tDCS decrease the excitability, in this study a constant current of 2 mA intensity was applied for 20 min.
  Arms: control; tDCS

SUMMARY:
Migraine has been described as one of the most common neurological diseases, with high social and economic impact. Despite the high prevalence, the pathophysiology of migraine is still unknown, several studies have been developed in order to advance the understanding of the pathophysiological mechanisms of the disease which are not yet entirely elucidated. The aim of this study is to observe the effects of transcranial direct current stimulation (tDCS), applied in the visual cortex, on neurophysiological and clinical measures (frequency, intensity, duration of attacks and severity of pain) in migraine patients.

ELIGIBILITY:
Inclusion criteria for migraine patients:

* Age must be between 18 to 40 years
* Gender: male and female
* Diagnosis must meet the 2004 IHS criteria for migraine without aura and migraine with aura
* Duration of the disease must be at least 12 months
* Patients had no preventative medication consistently for at least six months prior to study initiation.

Inclusion criteria for healthy individuals

* Age must be between 18 to 40 years
* Gender: male and female
* Individuals who have not filed headache crisis in the last year assessed according to the 2004 IHS criteria

Exclusion criteria

* Pregnant woman
* Individuals with clinical evidence of brain injury
* Metallic implant head
* Pacemaker
* History of seizure and chronic pain associated with other pathologies

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Change from phosphene threshold | At baseline,1 month, 2 months, 3 months/ per session - at baseline and 30 minutes (after tDCS)
  A 10-cm circular coil was used that has giving a peak magnetic field strength of 2 tesla. Subjects were asked to wear a blindfold, sit comfortably in a chair and to close their eyes to diminish ambient light.In sagittal line, three points were scored: 2, 3 and 4 cm above the inion. The single pulse transcranial magnetic stimulation was applied to one of the points scored and the subject was asked to report the presence or absence of a phosphene immediately after stimulation. The stimulation was repeated ten times at each intensity with a maximum frequency of 0.2 Hz, stimulation was initially applied to 60% of the maximum intensity of the stimulator. The intensity of stimulation was changed into blocks of 5% to minimum intensity that the subject can perceive the phosphene certainly, five times ten, then this value was set as the PT for migraineurs and controls.

SECONDARY OUTCOMES:
Change from eletroencephalography | At baseline, 1 month and 2 months, 3 months
  Electroencephalography was performed by digital EEG equipment, the sampling rate of 500 Hz, 0.5 Hz high pass filter and low pass 35 Hz to capture brain electrical activity through 23 electrodes on the scalp according to the International 10-20 system.After positioning the electrodes, the subject remained comfortably seated and relaxed, but awake, with eyes closed 30 cm from the photic stimulator and, without any stimulation, EEG was collected for 1 minute (baseline).After the baseline, was collected a sequence of 1 minute record without stimulation followed by 3 seconds to 9 Hz photic stimulation. This sequence is repeated 4 times. After this procedure, the subject received trains of visual stimuli, 20 seconds each, at frequencies of 3, 9, 15, 21 and 27 Hz, 1 minute spaced from each other and totaling 12 minutes evaluation.
Change from pain diary | 3 followed months
  The diary is a report of the frequency of the migraine attacks, the intensity, the onset and duration of the pain, the number of migraine-related days (the number of days on which the patients had migraine-related symptoms) and the type of analgesics in case of a migraine attack;

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Neuroscience Laboratory-LANA, Recife, Pernambuco, Brazil